CLINICAL TRIAL: NCT00338546
Title: Cocaine and Sympathetic Nerve Activity in Humans
Brief Title: Study to Improve Scientific Understanding of the Cardiovascular Actions of Cocaine
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2RO1DA01006409
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Cocaine Induced Sympathoexciation and Vasoconstriction
Keywords: Cocaine; Sympathetic nerve activity; Blood pressure; Cutaneous vasoconstriction; Coronary vasoconstriction
MeSH Terms: interventions — Cocaine; Dexmedetomidine; Laser-Doppler Flowmetry

INTERVENTIONS:
Drug: Cocaine hydrochloride
Drug: Dexmedetomidine
Procedure: Microneurography
Procedure: Laser doppler velocimetry

SUMMARY:
The purpose of this study is to improve the scientific understanding of the cardiovascular actions of cocaine, in particular the ability of cocaine to increase blood pressure.

DETAILED DESCRIPTION:
Cocaine abuse has emerged as a major cause of life-threatening cardiovascular emergencies but our understanding of the underlying mechanisms mediating the adverse effects of cocaine is far from complete. Our previous studies in cocaine-naive human subjects have demonstrated that intranasal cocaine acutely stimulates the human cardiovascular system by a novel central mechanism of action.We are currently investigating a central sympatholytic drug,dexmedetomidine, in reversing the sympathomimetic effects (increase in blood pressure, heart rate and coronary vasoconstriction) of intranasal cocaine.This drug may be a new pharmacologic agent in the treatment of acute cocaine intoxication in humans.

ELIGIBILITY:
Inclusion Criteria:

* Cocaine naive healthy volunteers

Exclusion Criteria:

* Any evidence of cardiopulmonary disease by history or physical examination
* History of hypertension or 24 hour blood pressure averaging >135/85 mmHg
* Any history of substance abuse (other than tobacco)
* Diabetes mellitus or other systemic illness
* Individuals with a history of pseudocholinesterase deficiency
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Blood pressure
Heart rate
Skin sympathetic nerve activity
Skin blood flow
Coronary blood flow

SECONDARY OUTCOMES:
Sedation status

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Victor, MD, Principal Investigator — Univ of Texas Southwestern Medical Center
Locations (1):
- Univ of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Result] Vongpatanasin W, Mansour Y, Chavoshan B, Arbique D, Victor RG. Cocaine stimulates the human cardiovascular system via a central mechanism of action. Circulation. 1999 Aug 3;100(5):497-502. doi: 10.1161/01.cir.100.5.497. PMID 10430763
- [Derived] Kontak AC, Victor RG, Vongpatanasin W. Dexmedetomidine as a novel countermeasure for cocaine-induced central sympathoexcitation in cocaine-addicted humans. Hypertension. 2013 Feb;61(2):388-94. doi: 10.1161/HYPERTENSIONAHA.112.203554. Epub 2013 Jan 2. PMID 23283356
- [Derived] Menon DV, Wang Z, Fadel PJ, Arbique D, Leonard D, Li JL, Victor RG, Vongpatanasin W. Central sympatholysis as a novel countermeasure for cocaine-induced sympathetic activation and vasoconstriction in humans. J Am Coll Cardiol. 2007 Aug 14;50(7):626-33. doi: 10.1016/j.jacc.2007.03.060. Epub 2007 Jul 30. PMID 17692748